CLINICAL TRIAL: NCT02503696
Title: Sample Collection Study to Evaluate DNA Markers in Subjects With Inflammatory Bowel Disease (IBD)
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2014-05
Record Dates: First submitted 2015-07-17; First posted 2015-07-21 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Inflammatory Bowel Disease; Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Colorectal Cancer
Keywords: Inflammatory Bowel Disease; Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Provide anonymous, clinically characterized specimens for bio-repository for future colorectal cancer-related test development.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD: Subjects will be men and women, 18-84 years of age, inclusive, who have been diagnosed with IBD. Each with a screening colonoscopy resulting in normal findings.
  Interventions: Device: Stool Collection Kit

INTERVENTIONS:
Device: Stool Collection Kit — Stool Collection Kit.

SUMMARY:
The primary objective of this study is to gather stool samples from subjects with inflammatory bowel disease (IBD) to be added to a test set of stool samples that will be utilized to help select molecular markers and determine the optimal sensitivity and specificity values for the Exact IBD-ACRN surveillance test for colorectal cancer (CRC).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18 - 84 years of age, inclusive, who have been diagnosed with IBD.
* Willing to provide a stool sample ≤120 but ≥7 days after a surveillance colonoscopy, which was negative for cancer/dysplasia.
* Written informed consent document signed and dated by the subject.

Exclusion Criteria:

* Any condition that in the opinion of the investigator should preclude participation in the study.
* A history of aerodigestive tract cancer.
* Prior colorectal resection, except ileocolic resection in Crohn's disease patients.
* IBD limited only to the rectum.
* Subject has participated in any clinical study within the previous 30 days wherein an investigational compound or device was, or may have been, introduced into the subject.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are at risk of developing colorectal cancer at the time of their colonoscopy and the colonoscopy resulted in normal findings.
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the Exact CRC diagnostic screening test. | 15 months
  The primary endpoint is point estimates of the sensitivity of the diagnostic test for detection of colorectal cancer in IBD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Lidgard, PhD, Study Chair — Exact Sciences
Locations (29):
- United States (27):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - UC San Diego Medical Center, La Jolla, California
  - Facey Medical Foundation, Mission Hills, California
  - Medical Research Center of Conneticut, Hamden, Connecticut
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, PC Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - HealthEast Midway Clinic, Saint Paul, Minnesota
  - Gastrointestinal Associates, Jackson, Mississippi
  - AGA Clinical Research Associates, LLC, Egg Harbor TWP, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - University of North Carolina, Chapel Hill, North Carolina
  - Kinston Medical Specialists, PA, Kinston, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - UC Health, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (2):
  - University of Calgary - Division of Gastroenterology, Calgary, Alberta
  - Winnipeg Regional Health Authority- Health Sciences, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No